CLINICAL TRIAL: NCT05278637
Title: DEVELOPMENT OF PROGNOSTIC PLATELET RNA BIOMARKERS TO TAILOR ANTIPLATELET THERAPY
Brief Title: GM03 - Platelet RNA Signatures of Aspirin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00048621
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Platelet Aggregation Inhibitors; Aspirin; Ticagrelor; RNA
MeSH Terms: interventions — Aspirin; Ticagrelor

STUDY DESIGN:
Intervention Model Description: 1. Aspirin 81mg/day x 4 weeks, Aspirin 325mg/day x 4 weeks, Aspirin washout, Ticagrelor 90mg BID x 4 weeks.
  2. Aspirin 325mg/day x 4 weeks, Aspirin 81mg/day x 4 weeks, Aspirin washout, Ticagrelor 90mg BID x 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aspirin 81mg/day, Aspirin 325mg/day, Aspirin washout, Ticagrelor 90mg BID (Active Comparator)
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Aspirin 325mg/day, Aspirin 81mg/day, Aspirin washout, Ticagrelor 90mg BID (Active Comparator)
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Ticagrelor 90mg BID (Active Comparator)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Aspirin — Aspirin 81mg/day x 4 weeks, Aspirin 325mg/day x 4 weeks. or Aspirin 325mg/day x 4 weeks, Aspirin 81mg/day x 4 weeks.
  Arms: Aspirin 325mg/day, Aspirin 81mg/day, Aspirin washout, Ticagrelor 90mg BID; Aspirin 81mg/day, Aspirin 325mg/day, Aspirin washout, Ticagrelor 90mg BID
Drug: Ticagrelor — Ticagrelor 90mg BID x 4 weeks

SUMMARY:
This study will involve healthy volunteers and patients with Type 2 diabetes. Eligible healthy volunteers will be invited to enroll into one of two protocols (A or B) and eligible patients with diabetes will be enrolled into protocol A.

DETAILED DESCRIPTION:
Protocol A This will be a randomized, cross-over design comparing low- and high-dose aspirin as well as a non-aspirin platelet inhibitor ticagrelor. This antiplatelet exposure study will be conducted at the DCRU using two separate cohorts: 1) healthy adult volunteers 2) patients with Type 2 diabetes. Subjects within each cohort will but in general will have platelet function testing and biospecimen collection before, four weeks, and eight weeks after low- or high-dose aspirin exposure. Subsequently there will be a period of aspirin washout and a four-week exposure to ticagrelor, a non-aspirin platelet inhibitor. In all subjects and at various time points peripheral blood RNA, purified platelets, DNA, serum, fecal samples and/or plasma will be collected.

Protocol B This will be a single arm study of the platelet inhibitor ticagrelor that is essentially the last two visits of Protocol A. This study will be conducted at the DCRU and will only be open to healthy adult volunteers and patients with Type 2 diabetes. Subjects who elect to participate in this protocol will follow the protocol outlined in Figure 2 and in general will have platelet function testing and biospecimen collection before and four weeks after exposure to ticagrelor, a non-aspirin platelet inhibitor. In all subjects and at various time points (see Figure 2 and Table 2) peripheral blood RNA, purified platelets, DNA, serum, and/ plasma will be collected. In order to align the visits with that of Protocol A, the two visits under this protocol will be labelled V4 and V5.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age ≥ 30 and ≤ 75
* Non-smoker
* The total number of enrolled females should not exceed 55% of the entire cohort. Therefore, the PI may include/exclude individuals on the basis of gender to achieve an equal balance between men and women.

Exclusion Criteria:

* History of bleeding disorder, gastrointestinal bleeding, intracranial bleeding or known prior gastric ulcer without documented resolution
* Current regular use of antiplatelet agents (aspirin, cilostazol, prasugrel, clopidogrel, dipyridamole, ticagrelor, or ticlopidine), nonsteroidal anti-inflammatory agents (NSAIDs), oral corticosteroids (i.e. prednisone), anticoagulants (warfarin, dabigatran, apixaban, rivaroxaban, enoxaparin)
* Known, severe hepatic impairment
* Surgery within the last 6 months, at the discretion of the PI
* Prior gastric bypass surgery (or equivalent) that interferes with absorbption at the discretion of the PI
* Aspirin allergy or known intolerance to aspirin or ticagrelor.
* Comorbid conditions:

  1. hypertension (requiring prescription medication).
  2. hyperlipidemia (requiring medications)
  3. Type 1 or 2 Diabetes

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

PRIMARY OUTCOMES:
Change in expression levels of platelet messenger RNA | Baseline, after every 4 week exposure

SECONDARY OUTCOMES:
Change in platelet function score | Baseline, 3 hours, after every 4 week exposure

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Voora, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No